CLINICAL TRIAL: NCT04189783
Title: Randomized Controlled Trial of Repeat vs. Single Quadratus Lumborum Block to Reduce Opioid Prescriptions After Open Resection of Retroperitoneal Sarcoma ("RESQU-SARC" Trial)
Brief Title: Repeat or Single Quadratus Lumborum Block for the Reduction of Opioid Prescriptions After Surgery in Retroperitoneal Sarcoma Patients ("RESQU-SARC" Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0780; NCI-2019-07564 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0780 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Retroperitoneal Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (liposomal bupivacaine) (Active Comparator): Patients receive standard of care liposomal bupivacaine injection before and during surgery and standard of care non-opioids and opioids at days 0-3 after surgery in the absence of unacceptable toxicity.
  Interventions: Drug: Liposomal Bupivacaine; Drug: Quadratus Lumborum Block; Other: Questionnaire Administration
- Arm II (liposomal bupivacaine) (Experimental): Patients receive standard of care liposomal bupivacaine injection before and during surgery and standard of care non-opioids and opioids at days 0-3 after surgery in the absence of unacceptable toxicity. Patients then receive a second liposomal bupivacaine injection on day 4 after surgery.
  Interventions: Drug: Liposomal Bupivacaine; Drug: Quadratus Lumborum Block; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Liposomal Bupivacaine — Patients receive standard of care liposomal bupivacaine injection before and during surgery, followed by standard of care non-opioids and opioids at days 0-3 after surgery in the absence of unacceptable toxicity
  Other Names: Bupivacaine Liposome Injectable Suspension; Exparel
Drug: Quadratus Lumborum Block — Patients receive standard of care liposomal bupivacaine injection before and during surgery, followed by standard of care non-opioids and opioids at days 0-3 after surgery in the absence of unacceptable toxicity. Patients receive a second liposomal bupivacaine injection ("RESQU" block) on day 4 after surgery
  Other Names: QL Block
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well a repeat or single liposomal bupivacaine injection (quadratus lumborum block) works in reducing opioid prescriptions after surgery in patients with retroperitoneal sarcoma. Liposomal bupivacaine is a numbing medication. Giving a second injection block may decrease dependency on opioid medications for pain relief after surgery and prevent long-term use and addiction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To use a pragmatic phase II randomized controlled trial to compare two standardized bundles of usual care for postoperative pain management to reduce the initial discharge prescription opioid volume.

SECONDARY OBJECTIVE:

I. To assess which pragmatic arm improves aspects of postoperative recovery including 30-day, 3-month, and 1-year opioid use, patient symptom inventory at those time points, hospital measures including length of stay and inpatient pain scores.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care liposomal bupivacaine injection before and during surgery and standard of care non-opioids and opioids at days 0-3 after surgery in the absence of unacceptable toxicity.

ARM II: Patients receive standard of care liposomal bupivacaine injection before and during surgery and standard of care non-opioids and opioids at days 0-3 after surgery in the absence of unacceptable toxicity. Patients then receive a second liposomal bupivacaine injection on day 4 after surgery.

After completion of study treatment, patients are followed up at 1, 3, and 12 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective open sarcoma resection for potentially curative intent who would otherwise be treated with quadratus lumborum (QL) block + intravenous-patient controlled analgesia (IV-PCA) converted to oral pain medications (meds) (non-narcotic bundle + opioid pain pill)

Exclusion Criteria:

* Patients with current or past substance (drug or alcohol) abuse disorder
* Laparoscopic or minimally invasive surgery
* Cases in which anticipated discharge is on or before postoperative day 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Scally, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 patients underwent resection, with 43 Arm-1 (Usual care) patients and 41 Arm-2 (2nd QL-block).
Pre-assignment Details: 29 participants were excluded from the study before assignment to arms due to screen failure, aborted surgery, discharged before 4 days after surgery or opioids free at 3rd day after surgery.
Groups:
- Arm 1, Control Arm (Usual Care): Arm 1 was a novel bundle (single block, 3 non-opioids, 5x-multiplier).
- Arm 2, Experimental Arm (2nd QL-Block): Arm 2 was the Arm 1 plus 2nd QL-block on POD4
Period: Overall Study
Arm/Group | Arm 1, Control Arm (Usual Care) | Arm 2, Experimental Arm (2nd QL-Block)
Started | 43 | 41
Completed | 43 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1, Control Arm (Usual Care) | Arm 2, Experimental Arm (2nd QL-Block) | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13.3) | 60 (12.7) | 58 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 28 | 24 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 36 | 34 | 70
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 37 | 36 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 43 | 41 | 84

OUTCOME MEASURES:

1. Primary Outcome: Initial Discharge Prescription Oral Morphine Equivalents (OME)
Description: After sarcoma surgery, our historical discharge opioid prescription was a median of 300mg oral morphine equivalents (OME) in 2016-2018, with 5% patients discharged opioid-free. The primary objective of this study was to compare 2 novel opioid-reduction bundles to increase the proportion of opioid-free patients.
Time Frame: At time of discharge (median of 9 days)
Measure: Median (Standard Deviation); unit: mg of Oral Morphine Equivalents (OME)
Arm/Group | Arm 1, Control Arm (Usual Care) | Arm 2, Experimental Arm (2nd QL-Block)
Number analyzed (Participants) | 43 | 41
mg of Oral Morphine Equivalents (OME) | 50 (444) | 25 (342)

2. Secondary Outcome: Proportion of Participants With Discharge Prescription OME = Zero
Description: Comparing the rate of opioid free patients at discharge between the 2 Arms
Time Frame: At time of discharge (median of 9 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Control Arm (Usual Care) | Arm 2, Experimental Arm (2nd QL-Block)
Number analyzed (Participants) | 43 | 41
Participants | 14 | 19

3. Secondary Outcome: Participant Reported Outcomes for Gastrointestinal Surgery- MD Anderson Symptom Inventory (MDASI-GI) at Discharge and 1 Month After Surgery.
Description: Compare the scores based on MDASI-GI between the 2 Arms. Score from 0 to 10 to define participant feelings with 0 for none and 10 for worst.
Time Frame: Scores at discharge and 1 month after the surgery
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1, Control Arm (Usual Care) | Arm 2, Experimental Arm (2nd QL-Block)
Number analyzed (Participants) | 43 | 41
score on a scale
  Pain score at discharge | 5 (3) | 4 (2)
  Pain score at 1 month | 3 (2) | 3 (3)
  General activity interference at discharge | 5 (3) | 4 (3)
  General activity interference at 1 month | 3 (2) | 3 (3)
  Interference with enjoyment of life at discharge | 4 (3) | 3 (3)
  Interference with enjoyment of life at 1 month | 2 (2) | 3 (3)

ADVERSE EVENTS:
Time Frame: Approximately 3 years, 5 months
Description: All surgical complications for 90 days after the surgery were recorded. They were all unrelated to the QL-Block. Eight patients died during the study, and they were all unrelated to the QL-Block.
Arm/Group | Arm 1, Control Arm (Usual Care) | Arm 2, Experimental Arm (2nd QL-Block)
All-Cause Mortality (participants affected / at risk) | 6/43 | 2/41
Serious Adverse Events (participants affected / at risk) | 9/43 | 10/41
Other Adverse Events (participants affected / at risk) | 6/43 | 7/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1, Control Arm (Usual Care) (N=43) | Arm 2, Experimental Arm (2nd QL-Block) (N=41)
Anemia requiring transfusion (Blood and lymphatic system disorders) | 0 | 1
Bladder leak requiring drain placement (Renal and urinary disorders) | 1 | 0
Delayed gastric emptying requiring percutaneous gastrostomy tube (Gastrointestinal disorders) | 0 | 1
Diarrhea requiring readmission (Gastrointestinal disorders) | 1 | 0
Intra-abdominal abscess/sepsis requiring emergent reoperation (Infections and infestations) | 0 | 1
Pancreatic leak requiring drainage (Hepatobiliary disorders) | 1 | 0
Pancreatic leak requiring IR drain (Hepatobiliary disorders) | 1 | 0
Partial small bowel obstruction (Gastrointestinal disorders) | 0 | 1
Pleural effusin (Gastrointestinal disorders) | 1 | 0
Postoperative hemorrhage requiring reintervention (Blood and lymphatic system disorders) | 1 | 0
Postoperative infection requiring re-intervention (Infections and infestations) | 0 | 2
Postoperative small bowel obstruction (Gastrointestinal disorders) | 0 | 1
Renal Obstruction requiring percutaneous nephrostomy (Renal and urinary disorders) | 1 | 0
Small bowel obstruction; intra-abdominal abscess (Gastrointestinal disorders) | 0 | 1
Ureteral obstruction requiring stent placement (Renal and urinary disorders) | 2 | 0
UTI treated with antibiotics (Infections and infestations) | 0 | 1
Wound dehiscence requiring repeat operation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1, Control Arm (Usual Care) (N=43) | Arm 2, Experimental Arm (2nd QL-Block) (N=41)
AKI (Renal and urinary disorders) | 0 | 1
Chyle leak requiring JP drain (Blood and lymphatic system disorders) | 1 | 0
Constipation, resolved w miralax (Gastrointestinal disorders) | 0 | 1
DVT treated with anticoagulation (General disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Prolonged ileus requiring NG placement and TPN (Gastrointestinal disorders) | 1 | 0
SSI requiring wound vac therapy (Infections and infestations) | 0 | 1
SSI, resolved w keflex (Infections and infestations) | 1 | 1
Superficial surgical infection (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
UTI treated with antibiotics (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT04189783/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT04189783/ICF_000.pdf